CLINICAL TRIAL: NCT04371029
Title: Impact of Neck Inspiratory Muscle Activation During Sleep in ICU Patients After a COVID 19 ARDS
Acronym: COVISLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2020/14
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: ARDS; COVID-19
Keywords: Neck inspiratory muscle (=NIM); Sleep; Intensive care unit; ARDS
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): A Polysomnography (PSG) will be performed in all patient the night before extubation, the day prior discharge and 3 month after. Recording will consist in EEG, EOG et EMG of the chin. We will record NIM EMG. We will also performed an actimetry during hospitalization in the post ICU ward. A quality of sleep questionnaire (Pittsburgh questionnaire) will be completed by the patients during the visit at 3 month.
  Interventions: Other: PSG

INTERVENTIONS:
Other: PSG — Polysomnography at 3 times, actimetry measure and Pittsburgh questionnaire

SUMMARY:
Most patients in intensive care units (ICUs) experience severe sleep disruption. Sleep disruption and sleep alteration may have an influence on the ability to breathe spontaneously. But, the cause of altered sleep remains unknown. Previous studies have shown that decreasing nocturnal respiratory muscle activity through mechanical ventilation might improve sleep quality. Nocturnal respiratory muscle activity may be one of the potential factor which contribute to alter sleep in the ICU. Therefore, the aim of this study is to analyse the presence of NIM activation during the night and it's consequence in an ICU population with the same pathology (COVID 19 ARDS).

DETAILED DESCRIPTION:
Sleep alteration is a common problem among ventilated ICU patient. About one third of the patient have abnormal EEG pattern which cannot be scored by using the AASM standard criteria. Patients experience marked fragmentation, absence of deep sleep, and REM sleep is decreased, . It has been shown that sleep deprivation has a negative impact on respiratory muscle endurance. So a good sleep is essential when the respiratory system is being challenged, as in the ICU during the weaning period. Indeed, in the ICU, patients with altered sleep, had a markedly longer weaning duration than in patients with normal sleep, and are more likely to fail a spontaneous breathing trial. Many factors may influence the quality of sleep in the ICU (noise, medication, mechanical ventilation …) but few studies have focus on the cause of this altered sleep, and the cause of altered sleep remains unknown. Previous studies have shown that decreasing nocturnal respiratory muscle activity through mechanical ventilation might improve sleep quality. Mechanical ventilation can decrease the charge imposed on the respiratory pump, and allows muscle to rest. Indeed, when the charge is too high (for example after an ARDS during the weaning period), the diaphragm may be overloaded, and there could be a greater involvement of other inspiratory muscles in breathing. In other pathological condition, the neck inspiratory muscle activity is increased (e.g. COPD, amyotrophic lateral sclerosis), and sometimes this activity persist during sleep with marked degradation in sleep architecture. Nocturnal respiratory muscle activity may be one of the potential factor which contribute to alter sleep in the ICU. Ttherefore, the aim of tis study is to analyse the presence of NIM activation during the night and it's consequence in an ICU population with the same pathology (COVID 19 ARDS).

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 year-old admitted to intensive care unit
* COVID-19 assessed by PCR on nasopharyngeal swab or pulmonary sample
* Oro-tracheal intubation for mechanical ventilation

Exclusion Criteria:

* Guardianship or curatorship
* Prisoners
* No health insurance
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with altered spleep | At day 10 after inclusion
  Comparison between patients with NIM activation during the night and patients without NIM activation during the night, in patients COVID 19 ARDS with altered spleep. A Polysomnography (PSG) will be performed the night before extubation.

SECONDARY OUTCOMES:
Sleep architecture at hospital discharge | At day 28 after inclusion
  Thanks to a PSG the night befor discharge, the seep architecture will be estimated.
Sleep monitoring during hospital stay after ICU discharge | At day 18 after ICU discharge
  Thanks to actimetry measure during hospitalization in the post ICU ward.
Sleep quality | 3 months after hospiotal discharge
  Sleep quality will be evaluate by the Pittsburgh sleep quality index. The 7 components of the score add up for give an overall score ranging from 0 to 21 points, 0 meaning that there is no difficulty, and 21 indicating on the contrary major difficulties.
Sleep architecture at month-3 | 3 months after hospital discharge
  Thanks to a PSG at 3 months, the seep architecture will be estimated.
Cost of ICU hospitalization | From inclusion to ICU discharge, up to 10 days after inclusion
  all cost will be estimated during ICU hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No